CLINICAL TRIAL: NCT02358733
Title: Use of Intra-Cytoplasmic Morphologically Selected Sperm Injection (IMSI) in Poor Responders to In Vitro Fertilization (IVF): a Prospective, Double-blind, Randomized, Controlled Trial
Brief Title: Use of IMSI in Poor Responders to IVF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DIfficulties with recruitment
Sponsor: Centro de Infertilidad y Reproducción Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRH-BROIMSI-2014; 2014-003928-50 (EudraCT Number)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Female Infertility
Keywords: POR; IMSI
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Intra-cytoplasmic Morphologically-selected Sperm Injection (IMSI)
  Interventions: Procedure: Intra-cytoplasmic Morphologically-selected Sperm Injection
- Control (Active Comparator): Intracytoplasmic sperm injection (ICSI)
  Interventions: Procedure: Intra-cytoplasmic Sperm Injection

INTERVENTIONS:
Procedure: Intra-cytoplasmic Sperm Injection — Selection of sperm at 400x for sperm injection
  Arms: Control
Procedure: Intra-cytoplasmic Morphologically-selected Sperm Injection — Selection of sperm at 6000x for sperm injection
  Arms: Treatment

SUMMARY:
This is a pilot study which aims to determine the role of IMSI in poor responders.

DETAILED DESCRIPTION:
This is a pilot study which aims to determine the role of IMSI over ICSI in poor responders to IVF, without a background of teratozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* poor ovarian response

Exclusion Criteria:

* body mass index (BMI) ≥ 30 kg/m2
* presence of endocrinopathies (e.g., diabetes, hyperprolactinemia, hypothyroidism)
* altered karyotype or documented genetic defects in one or both partners
* history of chronic, autoimmune or metabolic diseases
* altered meiosis in testicular biopsy or altered sperm-FISH
* teratozoospermia
* participation, simultaneously or within the previous 6 months, in another clinical trial with medication

Ages: 37 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2018-01 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Four to six weeks after embryo transfer
  Percentage of patients presenting with presence of an intrauterine gestational sac with embryonic cardiac activity display, evaluated by ultrasound, per cycle initiated

SECONDARY OUTCOMES:
Number of embryos obtained | Two days after egg retrieval
  Total number of embryos obtained
Percentage of cycles with embryo transfer | Two days after egg retrieval
  Number of cycles reaching embryo transfer per cycle initiated

CONTACTS AND LOCATIONS:
Overall Officials: Karinna Lattes, MD, Principal Investigator — Centro de Infertilidad y Reproducción Humana (CIRH)
Locations (1):
- Centro de Infertilidad y Reproducción Humana (CIRH), Barcelona, Spain